CLINICAL TRIAL: NCT05406076
Title: A Multicenter Randomized Controlled Study of the Efficacy of Oral Motor Therapy in Children With Autism
Brief Title: the Efficacy of Oral Motor Therapy in Children With Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Collaborators: Hefei Kanghua Rehabilitation Hospital (Unknown); Hefei Jingu Rehabilitation Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WDX-05
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-05

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Motor Therapy/ABA (Active Comparator): Eighty subjects who met the inclusion/exclusion criteria were randomly divided into 2 groups according to a 1:1 ratio. The experimental group was first treated with 2 months of ABA + oral motor therapy, followed by 2 months of ABA treatment.
  Oral motor therapy appliances can be used during mouth muscle training sessions, depending on the individual needs of the child. 30-40 min/session, 1 session/day, 5 sessions/week.
  ABA training time is at least 20 hours per week. The therapist is fully aware of each stage of the child's training during the teaching process and can make an accurate assessment of the child.
  Interventions: Behavioral: oral motor therapy; Behavioral: ABA
- ABA/Oral Motor Therapy (Active Comparator): Eighty subjects who met the inclusion/exclusion criteria were randomly divided into 2 groups according to a 1:1 ratio. The control group was treated with 2 months of ABA followed by 2 months of ABA + oral motor therapy.
  Oral motor therapy appliances can be used during mouth muscle training sessions, depending on the individual needs of the child. 30-40 min/session, 1 session/day, 5 sessions/week.
  ABA training time is at least 20 hours per week. The therapist is fully aware of each stage of the child's training during the teaching process and can make an accurate assessment of the child.
  Interventions: Behavioral: oral motor therapy; Behavioral: ABA

INTERVENTIONS:
Behavioral: oral motor therapy — Rigorous Chinese language oral motor therapy, including treatment of oral perceptual disorders and treatment of oral motor disorders. The treatment follows three basic principles: a combination of basic training and specific treatment; a combination of self-help and assisted treatment; and a combination of exercises, cues, and stimulation techniques. 30-40 min/session, 1 session/day, 5 sessions/week.
Behavioral: ABA — The mainstream ASD intervention approach with evidence-based support is currently recognized worldwide. Treatment follows the operational core principles of ABA, which are to establish learning goals based on the child's ability level, design teaching situations and select reinforcers for them, change the child's behavior problems with operational constraints, and to eliminate or improve problem behaviors through appropriate interventions to shape new adaptive behaviors. The training time is at least 20 hours per week.

SUMMARY:
Children with Autism spectrum disorders have speech disorders, which in turn aggravate communication difficulties and lead to an increase in their core symptoms. This experiment attempts to investigate the efficacy of Chinese language oral motor therapy in improving various aspects of articulation, language ability, and behavior of children with autism in conjunction with the International General Autism Scale, and provides a basis for the rational formulation of clinical treatment plans.

DETAILED DESCRIPTION:
Oral Motor Therapy (OMT) is a treatment process that uses tactile and proprioceptive stimulation techniques to promote the normalization of the sensory perception of the mouth (jaw, lips, tongue), suppress abnormal mouth movement patterns, and establish normal mouth movement patterns, following the principles of motor skill development.

This study investigates the efficacy of Chinese language oral motor therapy on improving various aspects of articulation, language ability, and behavior of children with autism. The study is divided into two parts, each eight weeks long. Eighty subjects who met the inclusion/exclusion criteria were randomly divided into 2 groups: the experimental group and the control group, in a 1:1 ratio. The experimental group was treated with 2 months of ABA+oral motor therapy followed by 2 months of ABA therapy; the control group was treated with 2 months of ABA therapy followed by 2 months of ABA+oral motor therapy.

Each subject underwent ABC, CARS, S-S, VB-MAPP, and ABLLS-R assessments before enrollment, 2 months after enrollment, and after discharge from the group.

ELIGIBILITY:
Inclusion Criteria:

1. Children who meet the DSM-V diagnosis of autism.
2. Age 2-5 years old, regardless of gender.
3. Native Chinese language.
4. No prior oral motor therapy.
5. Family members voluntarily participated in this study and signed an informed consent form.

Exclusion Criteria:

1. Children with co-occurring epilepsy.
2. Children with comorbid other psychiatric disorders.
3. Children with severe hearing impairment, history of visual impairment/blindness, organic disease of the mouth/throat, or significant medical illness or condition that prevents the child from participating in treatment procedures.
4. Children who received other oral motor training or speech articulation therapy during the intervention period.
5. Those who could not perform the intervention as planned after participating in the experiment.
6. Those deemed unsuitable by the investigator to participate in this experiment.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Verbal Behavior Milestones Assessment and Placement Program (VB-MAPP) scores | Baseline (week 0), Week 8，Week 16
  VB-MAPP is a criterion-referenced language and academic proficiency assessment system, curriculum instruction and skill tracking system for children with autism and speech and language delays. It is used for children 0-48 months of age. It has five components: milestone assessment, impairment assessment, transition assessment, task analysis, and supportive competencies and goals for placement and individualized education program (IEP).
Changes in Assessment of Basic Language and Learning Skills-Revised (ABLLS-R) scores | Baseline (week 0), Week 8，Week 16
  The ABLLS-R is for children ages 0-12. The scale has 25 major assessment items and 544 skill subtests that help children with autism learn the skills they need to communicate effectively and daily; and it can track the learning of each skill, which means that multiple assessments can be made, with the later assessment building on the previous one, giving this autism assessment tool a curriculum guide role.
Change in the Autism Behavior Scale (ABC) scores | Baseline (week 0), Week 8，Week 16
  The ABC scale is widely used in the assessment of autism conditions and the evaluation of treatment outcomes, and is one of the most commonly used autism assessment scales. It is used for screening of autistic individuals aged 18 months to 35 years. The scale is assessed by the child's parents or someone with whom the child has lived for at least 2 weeks and takes approximately 10-15 minutes to assess.
Change in Childhood Autism Rating Scale (CARS) scores | Baseline (week 0), Week 8，Week 16
  CARS is an observation tool used by clinicians for speech, behavior, and sensory perception in children with autism.
Change in China Rehabilitation Research Center version of the Sign-Significance（S-S，CRRC version） scores | Baseline (week 0), Week 8，Week 16
  The S-S detects the gap between the level of language delay and the actual age, as well as the status of the language delay, and is suitable for children aged 1-6.5 years with language delay. The test is administered individually and takes approximately 40 minutes to complete.